CLINICAL TRIAL: NCT00737386
Title: Frequency of Parasite Infection in Hyraxes and Sandflies During Outbreak of Leishmania Tropica Epidemic in The West Bank
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: David Enk, Professor, Hadassah Medical Organization
Other Study IDs: leishpeduel-HMO-CTIL
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmania tropica; Hyrax; Sandfly
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the project is to study the pathogenesis of Leishmania tropica infection in a focus of infection, to learn about relationship of infection in humans with ecological factors such as infection in hyraxes reservoir hosts and vector sandflies

ELIGIBILITY:
Inclusion Criteria:

* People living on regular basis in Peduel (the site of current leishmania tropica epidemic)with and without cutaneous signs of leishmania infection

Exclusion Criteria:

* None

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People living on regullar basis in Peduel (the site of current leishmania tropica epidemic)with and without cutaneous signs of leishmania infection
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel